CLINICAL TRIAL: NCT02187081
Title: Radiofrequency Ablation Accompanied With Spontaneous Sorafenib Administration in the Treatment of Early to Intermediate Stage Hepatocellular Carcinoma: a Prospective Multicenter Cohort Study.(REASSESS)
Brief Title: Radiofrequency Ablation Accompanied With Spontaneous Sorafenib in Early to Intermediate Stage HCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, feng xiaobin, Dr Xiaobin Feng, Southwest Hospital, China
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SWHB008
Record Dates: First submitted 2014-07-01; First posted 2014-07-10 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: HCC
Keywords: HCC; RFA; Sorafenib; Tumor recurrence; Overall survival
MeSH Terms: conditions — Recurrence | interventions — Radiofrequency Ablation; Sorafenib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sorafenib+RFA (Experimental): We give radiofrequency ablation plus Sorafenib for the treatment of HCC
  Interventions: Procedure: radiofrequency ablation plus Sorafenib
- RFA alone (Active Comparator): We give Radiofrequency ablation alone for the treatment of HCC
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: radiofrequency ablation plus Sorafenib — To treat HCC with the combination of radiofrequency ablation and sorafenib
  Arms: Sorafenib+RFA
Procedure: Radiofrequency ablation — To treat HCC with radiofrequency ablation alone.
  Arms: RFA alone

SUMMARY:
Radiofrequency ablation (RFA)can be curative with small localized HCCs up to 5 cm in diameter. However, the long-term prognosis is not satisfactory due to the high incidence of recurrence.Multimodality treatments are needed to prevent recurrences，but only useful with locoregional disease. Sorafenib is an oral multi-kinase inhibitor and the only systemic drug associated with improved overall survival (OS) in patients with advanced HCC. Retrospective and randomized studies have suggested that the combined use of Sorafenib may be useful in patients with unresectable HCC. Based on these information and the multiple actions of Sorafenib, we hypothesized that Sorafenib plus RFA may be useful in patients with early to Mid term HCC. In this investigation, we evaluated the safety and efficacy of a combination Sorafenib and RFA therapy in patients with Barcelona Clinic Liver Cancer (BCLC) Stage 0 -B1 HCC in a multicenter prospective cohort study.

DETAILED DESCRIPTION:
Radiofrequency ablation (RFA) has been used as a minimally invasive option to eradicate tumors and preserve liver function in patients with impaired function or with a postoperative tumor recurrence. RFA can be curative with small localized HCCs up to 5 cm in diameter. However, the long-term prognosis for HCC patients treated with RFA is not satisfactory due to the high incidence of recurrence including local tumor recurrence and multicentric carcinogenesis.

Multimodality treatments are needed to prevent recurrences. Although there is a potential benefit with this strategy, it is only useful with locoregional disease. Sorafenib is an oral multi-kinase inhibitor and the only systemic drug associated with improved overall survival (OS) in patients with advanced HCC.

Retrospective and randomized studies have suggested that the combined use of Sorafenib, TACE, and RFA may be useful in patients with unresectable HCC. Based on these information and the multiple actions of Sorafenib, we hypothesized that Sorafenib plus RFA may be useful in patients with early HCC or recurrent HCC. Although no supportive data from clinical trials is available, this hypothesis is supported by recent animal studies. Inadequate RFA has been shown to promote rapid progression of residual tumors. Adjuvant Sorafenib postponed time to recurrence by inhibition of hypoxia inducible factor-1and vascular endothelial growth factor A (VEGFA). In a multifocal tumor model of HCC, RFA and Sorafenib alone resulted in a significant volume reduction of non-RFA-targeted tumors, but this effect was enhanced when both modalities were combined. This phenomenon was also demonstrated by more recent study on human subject.

Besides the advantages, Sorafenib initially promoted necrosis, delayed tissue repair after RFA and adversely affected normal liver parenchyma, which could result in increased RFA toxicity and limit its use in patients with HCC who have undergone RFA. Thus, the overall advantages of RFA plus Sorafenib need to be weighed against its adverse effects. In this investigation, we evaluated the safety and efficacy of a combination Sorafenib and RFA therapy in patients with Barcelona Clinic Liver Cancer (BCLC) Stage 0 -B1 HCC in a multicenter prospective cohort study.

Outcome measures: Post-RFA tumor recurrence

ELIGIBILITY:
Inclusion Criteria:

* Authorization of Informed Consent
* HCC diagnosed by biopsy or Image findings
* BCLC stage 0 to B1
* This time was the primary treatment of HCC. Had no history of any tumor specific therapy,including RFA,Hepatectomy,TACE,HIFU,and Transplantation
* Child Pugh A or B
* ECOG 0 to 2
* single lesion less than or equal to 5 cm,2 to 3 nodules, maximal size less than equal to 3cm
* Male or female (without pregnancy)
* Ages between 18 to 70 years
* Capable of take medicines
* anticipate at least survival of 12 weeks
* Unwilling to receive surgical resection or liver transplantation
* Potentially curable disease by RFA
* Sorafenib administrated less than 4 weeks before or after RFA procedures
* For any excuse,subject should take Sorafenib at least for 4 weeks

Exclusion Criteria:

* A cancer embolus in major hepatic vessels or extrahepatic metastases
* Tumor number more than 4 or tumor size larger than 5 cm
* A present or past history of uncontrollable ascites, hepatic encephalopathy or variceal bleeding
* A history of a secondary malignancy
* Severe dysfunction of the heart, kidney or other organs
* Active infection except viral hepatitis
* Any treatment history of target lesion including chemotherapy and TACE
* Pregnancy
* received other trials on gene therapy
* have received operation less than 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
2-year incidence of tumor recurrence | 2 year
  to calculate the incidence of tumor recurrence of experiment and control group at two year after complete treatment.

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival
1-year incidence of recurrence | 1-year
  1-year incidence of recurrence
3-year incidence of recurrence | 3 year
  3-year incidence of recurrence
5-year incidence of recurrence | 5 year
  5-year incidence of recurrence
Time to progression | average 2 years
  Time to progression
Disease Control Rate | average 2 years
  Disease Control Rate
complications and adverse effect | 1 year
  to sum all the complications and adverse effect for all the eligible enrolled patients during 1 year of a complete treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China